CLINICAL TRIAL: NCT03992170
Title: A Pilot Study on the Efficacy of Daratumumab in Multiple Myeloma (MM) Patients in >VGPR/MRD-positive by Next Generation Flow
Brief Title: Study of Daratumumab in Multiple Myeloma (MM) Patients in >VGPR/MRD-positive
Acronym: DART4MM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Collaborators: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Principal Investigator, Alessandro Gozzetti, Professor, Azienda Ospedaliera Universitaria Senese
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DART4MM
Record Dates: First submitted 2019-06-03; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Myeloma Multiple
Keywords: Myeloma Multiple; Daratumumab
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Patients will receive Daratumumab (16 mg/Kg day) every week for 8 weeks intravenous (8 infusions) and then every 2 weeks for 16 weeks intravenous (8 more infusions).
  If MRD positive by NGF, the patients will receive Daratumumab every 4 weeks for 80 weeks intravenous; if MRD negative by NGF, the patients can stop the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Patients will receive Daratumumab (16 mg/Kg day) every week for 8 weeks intravenous (8 infusions) and then every 2 weeks for 16 weeks intravenous (8 more infusions).
  If MRD positive by NGF, the patients will receive Daratumumab every 4 weeks for 80 weeks intravenous; if MRD negative by NGF, the patients can stop the treatment.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab is a human monoclonal antibody (mAb) IgG1 that binds to the highly expressed CD38 protein on the surface of multiple myeloma cells and, at various levels, also in other types of cells and tissues. The CD38 protein has multiple functions, such as receptor-mediated adhesion, signal transduction activity and enzymatic activity.
  Other Names: Darzalex

SUMMARY:
Aim of this study is to evaluate Daratumumab effect on MRD-positive patients with Multiple Myeloma (MM) who achieved >VGPR after any therapy (ASCT, VMP, Rev-Dex). Daratumumab 16 mg/kg administered at weekly intervals for 8 weeks, then every 2 weeks for an additional 16 weeks, will be given to 50 MM patients who achieved a >VGPR defined by monoclonal component disappearance in serum or urine, immunofixation positive/negative and MRD-positivity (by NGF). Free light chain (FLC) and CT/PET will be evaluated at time 0. NGF will be done on marrow aspirate at time 0, at 2 months and every 6 months for 2 years. If patients will be still MRD positive after 6 months of therapy , treatment will be continued up to 2 years. If MRD negative by NGF, the patients can stop the treatment.

DETAILED DESCRIPTION:
Daratumumab in clinical trials and study rationale Daratumumab is an immunoglobulin G1 kappa (IgG1κ) human mAb against CD 38 antigen, produced in a mammalian cell line (CHO) using recombinant DNA technology. (see Investigational Brochure, IB) Daratumumab has been explored as a single agent in relapsed and refractory patients (GEN501,NCT00574288. In the dose-expansion phase 30 patients received 8 mg/kg and 42 patients 16 mg/kg once weekly (8 doses), twice monthly (8 doses) then monthly up to 24 months. Patients had received a median number of 4 to 5 lines of therapy with 54% of patients refractory to bortezomib and 72% to lenalidomide. Low grade infusion-related reactions were initially observed in up to 75% of patients but were considerably attenuated by the delivery in a large infusion volume. Thirty five percent of patients receiving a dose of 16 mg/kg responded, with 15% of complete or very good partial responses. These encouraging results were confirmed in the multicenter phase 2 study SIRIUS (NCT01985126). In this study, 106 heavily pretreated myeloma patients received daratumumab monotherapy (16 mg/kg). Patients had received a median of 5 prior therapies and the majority of them were refractory to bortezomib, lenalidomide and pomalidomide. Partial response was achieved by 29.2% of patients and the median duration of response was 7.4 months.

A pooled analysis of the patients of the GEN 501 and the SIRIUS trials who had received daratumumab monotherapy at the dose of 16 mg/kg (n=148) showed an overall response rate of 31.1% and a median PFS and OS of 4 and 20 months, respectively. Patients achieving only stable disease or minimal response reached a promising median overall survival of 18.5 months, which is unexpected in this population of very advanced myeloma patients. The quality of response was correlated with the expression intensity of CD38 by neoplastic plasmocytes. Daratumumab was granted accelerated approval in 2015 by the FDA to treat patients with multiple myeloma who had received at least three prior treatments. Daratumumab is also being studied in combination with many other agents including lenalidomide, bortezomib, carfilzomib or pomalidomide. The phase 3 randomized trial CASTOR recently confirmed a strong advantage of the addition of daratumumab to bortezomib/dexamethasone, in 498 relapsed myeloma patients (NCT02136134). The triplet combination was associated with a significantly better response rate, including 82.9% of PR or better and 19.2% of CR or better. The 1-year rate of progression free survival was 60.7% in the daratumumab group versus 26.9% in the control arm. The updated results of this trial have confirmed this strong PFS benefit for the patients in the daratumumab arm, especially for the patients in first relapse (12-months PFS : 77.3% vs 24.7%, p<10-4). Daratumumab also clearly improved the median PFS of patients with high-risk cytogenetic. In this relapse setting, the POLLUX trial also demonstrated a strong advantage of the addition of daratumumab to lenalidomide and dexamethasone, in terms of both response rate and PFS (NCT02076009) . In this trial, patients in the daratumumab group reached an overall response rate of 93% (including 43% CR) and had a 63% reduction in the risk of progression. The updated results of this trial confirmed this significant PFS advantage even in lenalidomide-naïve patients and in patients with high-risk cytogenetic. Minimal Residual disease (MRD) assessed by NGS analysis in patients included in CASTOR and POLLUX trials revealed an unprecedently observed rate of patients with MRD negative disease. Indeed, 32% (vs 9%) and 18% (vs 4%) of patients reached a 10-4 MRD negative in the daratumumab (versus control) arms of POLLUX and CASTOR, respectively. In particular the rate of MRD negativity (10-5) has increased continuosly after month 6 in patients receiving Daratumumab monotherapy in the CASTOR trial. (36) The addition of daratumumab is currently being assessed in the context of previously untreated myeloma patients. The phase 3 randomized study Cassiopeia is currently evaluating the role of daratumumab in combination with VTD in induction, and its role as maintenance after high-dose therapy (NCT02541383). In patients not eligible for transplant, the phase 3 randomized trial MAIA is evaluating the addition of daratumumab to lenalidomide-dexamethasone (NCT02252172). In the ALCYONE trial (Dara-VMP vs VMP) in patients inelegible to transplant MRD negativity (10-5) has increased continuosly after cycle 10 with daratumumab monotherapy.(37) The potential benefit of daratumumab has also been recently evaluated in high-risk smoldering myeloma patients in the phase 3 randomized CENTAURUS (NCT02316106). Daratumumab monotherapy can increase response and in particular MRD negativity, which correlates with PFS and OS. To the investigator's knowledge the use of daratumumab in multiple myeloma patients with suboptimal response (in particular with a >VGPR/MRD+) has not yet been explored. To achieve a better response can ameliorate patient outcome and survival.

DATA COLLECTION All patient-related data are recorded in a pseudonomized way. Each patient is unequivocally identified by a trial subject number, attributed at recruitment into the study. The investigator has to keep a patient identification log, including the full name and address of the subject and eventually additional relevant personal data such as hospital record number, home physician etc. In addition, patients who were screened in order to be entered into the study, but who could not be recruited for whatever reason (informed consent not given, not fulfilling selection criteria etc.) are recorded in a "patient reject log". All the data retrieved during the conduct of the study are entered into the appropriate case record forms (CRF) by the investigator or another person authorized by the investigator (co-investigator). The CRFs are provided by the study secretariat and are explained to the investigator by the study monitor.

SAMPLE SIZE CALCULATION The main objective of the trial is to assess, whether the experimental regimen shows a promising activity profile in treatment of MM minimal residual disease. The primary endpoint is the response rate. Multiple myeloma patients achieving CR and MRD negativity after autotransplant are around 60% and 20% of the total, respectively. MM patients that achieve an MRD negative status after VMP (velcade , melphalan prednisone) are not known. Since CR achievement after VMP is 30%, MRD negativity is probably < 5% of the patients. Statistical analysis will be provided on 50 patients, assuming the power to show an increase in MRD negativity from 20% to at least 50% of the patients treated. In summary, the trial design is based on the following assumptions: The activity of the experimental therapy would be rated as insufficient, if the actual response rate was only 20% or lower. On the other hand, the regimen would be considered to be a promising candidate for further development (e.g. in a phase III trial), if the true ORR amounted to 50% or more. To show effectiveness of daratumumab to give a negative MRD; only descriptive statistics will be performed AE RECORDING All adverse events and special reporting situations, whether serious or non-serious, will be reported from the time a signed and dated ICF is obtained until completion of the subject's last study-related procedure, which may include contact for follow-up of safety. Serious adverse events, including those spontaneously reported to the investigator within 30 days after the last dose of study drug, must be reported using the Serious Adverse Event Form. The sponsor will evaluate any safety information that is spontaneously reported by an investigator beyond the time frame specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Able to adhere to the study visit schedule and other protocol requirements
* >VGPR/MRD-positive by NGF measured by 2-tubes optimized 8-color antibody panel, (OneFlow PCST e PCD BD Biosciences)
* Patients should be at enrollment at least 12 weeks from any therapy for myeloma after diagnosis or at any subsequent relapse
* Eastern Cooperative Oncology Group performance status score of 0, 1, or 2
* Laboratory values and electrocardiogram within protocol-defined parameters at screening
* All previous MM therapy, including radiation, cytostatic therapy and surgery, must have been terminated at least 4 weeks prior to treatment in this study, without corticosteroid therapy.
* Laboratory test results within these ranges:

  * Absolute neutrophil count 1.0 x 109/L
  * Platelet count 75 x 109/L
  * Creatinine clearance > 30 ml/h)
  * Total bilirubin 1.5 mg/Dl
  * Aspartate aminotransferase (AST; SGOT) and alanine aminotransferase (ALT; SGPT) 2 x ULN
* Disease free of prior malignancies for 5 years with exception of curatively treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* Fertile patients must use effective contraception during and for 6 months after study treatment
* Patients must sign on an Informed Consent Form No study treatment or any other procedure within the framework of the trial (except for screening) will be performed in any patient prior to receipt of written informed consent.

Exclusion Criteria:

* Received Daratumumab or other anti-CD38 therapies previously
* Nonsecretory multiple myeloma
* Previously received an allogenic stem cell transplant or has received an autologous stem cell transplantation within 12 weeks
* Known chronic obstructive pulmonary disease, persistent asthma, or a history of asthma within 5 years
* Absence of the Informed Consent Form signed by the patient
* Pregnant or breast feeding females
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to the study drugs
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C.
* Plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or amyloidosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Responde Rate (ORR) | every 6 months
  The fraction of patients who experience a Minimal Residual Disease (MRD) negativity per IMWG 2016 criteria

SECONDARY OUTCOMES:
Progression free survival (PFS) | every 6 months
  PFS determined using the Kaplan-Meier method, considering those who progress or die without progression as failures, and censoring those who do not
Complete Remission Rate (CR) | every 6 months
  The fraction of patient who experience a sCR using the study treatment
Duration of Response (DoR) | every 6 months
  The fraction of patients who continues to respond to treatment without Myeloma progression

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Gozzetti, Medicine, Principal Investigator — Azienda Ospedaliera Universitaria Senese
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kyle RA, Rajkumar SV. Multiple myeloma. Blood. 2008 Mar 15;111(6):2962-72. doi: 10.1182/blood-2007-10-078022. PMID 18332230
- [Background] Brenner H, Gondos A, Pulte D. Recent major improvement in long-term survival of younger patients with multiple myeloma. Blood. 2008 Mar 1;111(5):2521-6. doi: 10.1182/blood-2007-08-104984. Epub 2007 Sep 27. PMID 17901246
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Background] Gozzetti A, Cerase A, Lotti F, Rossi D, Palumbo A, Petrucci MT, Patriarca F, Nozzoli C, Cavo M, Offidani M, Floridia M, Berretta S, Vallone R, Musto P, Lauria F; GIMEMA (Gruppo Italiano Malattie Ematologiche dell'Adulto) Myeloma Working Party; Marchini E, Fabbri A, Oliva S, Zamagni E, Sapienza FG, Ballanti S, Mele G, Galli M, Pirrotta MT, Di Raimondo F. Extramedullary intracranial localization of multiple myeloma and treatment with novel agents: a retrospective survey of 50 patients. Cancer. 2012 Mar 15;118(6):1574-84. doi: 10.1002/cncr.26447. Epub 2011 Aug 25. PMID 21932386
- [Background] Ocio EM, Richardson PG, Rajkumar SV, Palumbo A, Mateos MV, Orlowski R, Kumar S, Usmani S, Roodman D, Niesvizky R, Einsele H, Anderson KC, Dimopoulos MA, Avet-Loiseau H, Mellqvist UH, Turesson I, Merlini G, Schots R, McCarthy P, Bergsagel L, Chim CS, Lahuerta JJ, Shah J, Reiman A, Mikhael J, Zweegman S, Lonial S, Comenzo R, Chng WJ, Moreau P, Sonneveld P, Ludwig H, Durie BG, Miguel JF. New drugs and novel mechanisms of action in multiple myeloma in 2013: a report from the International Myeloma Working Group (IMWG). Leukemia. 2014 Mar;28(3):525-42. doi: 10.1038/leu.2013.350. Epub 2013 Nov 20. PMID 24253022
- [Background] Fonseca R, Blood E, Rue M, Harrington D, Oken MM, Kyle RA, Dewald GW, Van Ness B, Van Wier SA, Henderson KJ, Bailey RJ, Greipp PR. Clinical and biologic implications of recurrent genomic aberrations in myeloma. Blood. 2003 Jun 1;101(11):4569-75. doi: 10.1182/blood-2002-10-3017. Epub 2003 Feb 6. PMID 12576322
- [Background] Gozzetti A, Le Beau MM. Fluorescence in situ hybridization: uses and limitations. Semin Hematol. 2000 Oct;37(4):320-33. doi: 10.1016/s0037-1963(00)90013-1. PMID 11071355
- [Background] Stewart AK, Richardson PG, San-Miguel JF. How I treat multiple myeloma in younger patients. Blood. 2009 Dec 24;114(27):5436-43. doi: 10.1182/blood-2009-07-204651. Epub 2009 Oct 27. PMID 19861683
- [Background] Moreau P, Avet-Loiseau H, Harousseau JL, Attal M. Current trends in autologous stem-cell transplantation for myeloma in the era of novel therapies. J Clin Oncol. 2011 May 10;29(14):1898-906. doi: 10.1200/JCO.2010.32.5878. Epub 2011 Apr 11. PMID 21482979
- [Background] Harousseau JL, Attal M, Avet-Loiseau H, Marit G, Caillot D, Mohty M, Lenain P, Hulin C, Facon T, Casassus P, Michallet M, Maisonneuve H, Benboubker L, Maloisel F, Petillon MO, Webb I, Mathiot C, Moreau P. Bortezomib plus dexamethasone is superior to vincristine plus doxorubicin plus dexamethasone as induction treatment prior to autologous stem-cell transplantation in newly diagnosed multiple myeloma: results of the IFM 2005-01 phase III trial. J Clin Oncol. 2010 Oct 20;28(30):4621-9. doi: 10.1200/JCO.2009.27.9158. Epub 2010 Sep 7. PMID 20823406
- [Background] Cavo M, Tacchetti P, Patriarca F, Petrucci MT, Pantani L, Galli M, Di Raimondo F, Crippa C, Zamagni E, Palumbo A, Offidani M, Corradini P, Narni F, Spadano A, Pescosta N, Deliliers GL, Ledda A, Cellini C, Caravita T, Tosi P, Baccarani M; GIMEMA Italian Myeloma Network. Bortezomib with thalidomide plus dexamethasone compared with thalidomide plus dexamethasone as induction therapy before, and consolidation therapy after, double autologous stem-cell transplantation in newly diagnosed multiple myeloma: a randomised phase 3 study. Lancet. 2010 Dec 18;376(9758):2075-85. doi: 10.1016/S0140-6736(10)61424-9. Epub 2010 Dec 9. PMID 21146205
- [Background] Rosinol L, Oriol A, Teruel AI, Hernandez D, Lopez-Jimenez J, de la Rubia J, Granell M, Besalduch J, Palomera L, Gonzalez Y, Etxebeste MA, Diaz-Mediavilla J, Hernandez MT, de Arriba F, Gutierrez NC, Martin-Ramos ML, Cibeira MT, Mateos MV, Martinez J, Alegre A, Lahuerta JJ, San Miguel J, Blade J; Programa para el Estudio y la Terapeutica de las Hemopatias Malignas/Grupo Espanol de Mieloma (PETHEMA/GEM) group. Superiority of bortezomib, thalidomide, and dexamethasone (VTD) as induction pretransplantation therapy in multiple myeloma: a randomized phase 3 PETHEMA/GEM study. Blood. 2012 Aug 23;120(8):1589-96. doi: 10.1182/blood-2012-02-408922. Epub 2012 Jul 12. PMID 22791289
- [Background] Sonneveld P, Schmidt-Wolf IG, van der Holt B, El Jarari L, Bertsch U, Salwender H, Zweegman S, Vellenga E, Broyl A, Blau IW, Weisel KC, Wittebol S, Bos GM, Stevens-Kroef M, Scheid C, Pfreundschuh M, Hose D, Jauch A, van der Velde H, Raymakers R, Schaafsma MR, Kersten MJ, van Marwijk-Kooy M, Duehrsen U, Lindemann W, Wijermans PW, Lokhorst HM, Goldschmidt HM. Bortezomib induction and maintenance treatment in patients with newly diagnosed multiple myeloma: results of the randomized phase III HOVON-65/ GMMG-HD4 trial. J Clin Oncol. 2012 Aug 20;30(24):2946-55. doi: 10.1200/JCO.2011.39.6820. Epub 2012 Jul 16. PMID 22802322
- [Background] Richardson PG, Weller E, Lonial S, Jakubowiak AJ, Jagannath S, Raje NS, Avigan DE, Xie W, Ghobrial IM, Schlossman RL, Mazumder A, Munshi NC, Vesole DH, Joyce R, Kaufman JL, Doss D, Warren DL, Lunde LE, Kaster S, Delaney C, Hideshima T, Mitsiades CS, Knight R, Esseltine DL, Anderson KC. Lenalidomide, bortezomib, and dexamethasone combination therapy in patients with newly diagnosed multiple myeloma. Blood. 2010 Aug 5;116(5):679-86. doi: 10.1182/blood-2010-02-268862. Epub 2010 Apr 12. PMID 20385792
- [Background] Kumar S, Flinn I, Richardson PG, Hari P, Callander N, Noga SJ, Stewart AK, Turturro F, Rifkin R, Wolf J, Estevam J, Mulligan G, Shi H, Webb IJ, Rajkumar SV. Randomized, multicenter, phase 2 study (EVOLUTION) of combinations of bortezomib, dexamethasone, cyclophosphamide, and lenalidomide in previously untreated multiple myeloma. Blood. 2012 May 10;119(19):4375-82. doi: 10.1182/blood-2011-11-395749. Epub 2012 Mar 15. PMID 22422823
- [Background] Jakubowiak AJ, Dytfeld D, Griffith KA, Lebovic D, Vesole DH, Jagannath S, Al-Zoubi A, Anderson T, Nordgren B, Detweiler-Short K, Stockerl-Goldstein K, Ahmed A, Jobkar T, Durecki DE, McDonnell K, Mietzel M, Couriel D, Kaminski M, Vij R. A phase 1/2 study of carfilzomib in combination with lenalidomide and low-dose dexamethasone as a frontline treatment for multiple myeloma. Blood. 2012 Aug 30;120(9):1801-9. doi: 10.1182/blood-2012-04-422683. Epub 2012 Jun 4. PMID 22665938
- [Background] Sonneveld P, Asselbergs E, Zweegman S, van der Holt B, Kersten MJ, Vellenga E, van Marwijk-Kooy M, Broyl A, de Weerdt O, Lonergan S, Palumbo A, Lokhorst H. Phase 2 study of carfilzomib, thalidomide, and dexamethasone as induction/consolidation therapy for newly diagnosed multiple myeloma. Blood. 2015 Jan 15;125(3):449-56. doi: 10.1182/blood-2014-05-576256. Epub 2014 Nov 14. PMID 25398935
- [Background] Ladetto M, Pagliano G, Ferrero S, Cavallo F, Drandi D, Santo L, Crippa C, De Rosa L, Pregno P, Grasso M, Liberati AM, Caravita T, Pisani F, Guglielmelli T, Callea V, Musto P, Cangialosi C, Passera R, Boccadoro M, Palumbo A. Major tumor shrinking and persistent molecular remissions after consolidation with bortezomib, thalidomide, and dexamethasone in patients with autografted myeloma. J Clin Oncol. 2010 Apr 20;28(12):2077-84. doi: 10.1200/JCO.2009.23.7172. Epub 2010 Mar 22. PMID 20308672
- [Background] Cerrato C, Palumbo A. Initial treatment of nontransplant patients with multiple myeloma. Semin Oncol. 2013 Oct;40(5):577-84. doi: 10.1053/j.seminoncol.2013.07.003. PMID 24135402
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Gay F, Larocca A, Wijermans P, Cavallo F, Rossi D, Schaafsma R, Genuardi M, Romano A, Liberati AM, Siniscalchi A, Petrucci MT, Nozzoli C, Patriarca F, Offidani M, Ria R, Omede P, Bruno B, Passera R, Musto P, Boccadoro M, Sonneveld P, Palumbo A. Complete response correlates with long-term progression-free and overall survival in elderly myeloma treated with novel agents: analysis of 1175 patients. Blood. 2011 Mar 17;117(11):3025-31. doi: 10.1182/blood-2010-09-307645. Epub 2011 Jan 12. PMID 21228328
- [Background] Facon T, Mary JY, Hulin C, Benboubker L, Attal M, Pegourie B, Renaud M, Harousseau JL, Guillerm G, Chaleteix C, Dib M, Voillat L, Maisonneuve H, Troncy J, Dorvaux V, Monconduit M, Martin C, Casassus P, Jaubert J, Jardel H, Doyen C, Kolb B, Anglaret B, Grosbois B, Yakoub-Agha I, Mathiot C, Avet-Loiseau H; Intergroupe Francophone du Myelome. Melphalan and prednisone plus thalidomide versus melphalan and prednisone alone or reduced-intensity autologous stem cell transplantation in elderly patients with multiple myeloma (IFM 99-06): a randomised trial. Lancet. 2007 Oct 6;370(9594):1209-18. doi: 10.1016/S0140-6736(07)61537-2. PMID 17920916
- [Background] Palumbo A, Bringhen S, Caravita T, Merla E, Capparella V, Callea V, Cangialosi C, Grasso M, Rossini F, Galli M, Catalano L, Zamagni E, Petrucci MT, De Stefano V, Ceccarelli M, Ambrosini MT, Avonto I, Falco P, Ciccone G, Liberati AM, Musto P, Boccadoro M; Italian Multiple Myeloma Network, GIMEMA. Oral melphalan and prednisone chemotherapy plus thalidomide compared with melphalan and prednisone alone in elderly patients with multiple myeloma: randomised controlled trial. Lancet. 2006 Mar 11;367(9513):825-31. doi: 10.1016/S0140-6736(06)68338-4. PMID 16530576
- [Background] Palumbo A, Bringhen S, Liberati AM, Caravita T, Falcone A, Callea V, Montanaro M, Ria R, Capaldi A, Zambello R, Benevolo G, Derudas D, Dore F, Cavallo F, Gay F, Falco P, Ciccone G, Musto P, Cavo M, Boccadoro M. Oral melphalan, prednisone, and thalidomide in elderly patients with multiple myeloma: updated results of a randomized controlled trial. Blood. 2008 Oct 15;112(8):3107-14. doi: 10.1182/blood-2008-04-149427. Epub 2008 May 27. PMID 18505783
- [Background] Wijermans P, Schaafsma M, Termorshuizen F, Ammerlaan R, Wittebol S, Sinnige H, Zweegman S, van Marwijk Kooy M, van der Griend R, Lokhorst H, Sonneveld P; Dutch-Belgium Cooperative Group HOVON. Phase III study of the value of thalidomide added to melphalan plus prednisone in elderly patients with newly diagnosed multiple myeloma: the HOVON 49 Study. J Clin Oncol. 2010 Jul 1;28(19):3160-6. doi: 10.1200/JCO.2009.26.1610. Epub 2010 Jun 1. PMID 20516439
- [Background] Hulin C, Facon T, Rodon P, Pegourie B, Benboubker L, Doyen C, Dib M, Guillerm G, Salles B, Eschard JP, Lenain P, Casassus P, Azais I, Decaux O, Garderet L, Mathiot C, Fontan J, Lafon I, Virion JM, Moreau P. Efficacy of melphalan and prednisone plus thalidomide in patients older than 75 years with newly diagnosed multiple myeloma: IFM 01/01 trial. J Clin Oncol. 2009 Aug 1;27(22):3664-70. doi: 10.1200/JCO.2008.21.0948. Epub 2009 May 18. PMID 19451428
- [Background] Waage A, Gimsing P, Fayers P, Abildgaard N, Ahlberg L, Bjorkstrand B, Carlson K, Dahl IM, Forsberg K, Gulbrandsen N, Haukas E, Hjertner O, Hjorth M, Karlsson T, Knudsen LM, Nielsen JL, Linder O, Mellqvist UH, Nesthus I, Rolke J, Strandberg M, Sorbo JH, Wisloff F, Juliusson G, Turesson I; Nordic Myeloma Study Group. Melphalan and prednisone plus thalidomide or placebo in elderly patients with multiple myeloma. Blood. 2010 Sep 2;116(9):1405-12. doi: 10.1182/blood-2009-08-237974. Epub 2010 May 6. PMID 20448107
- [Background] Beksac M, Haznedar R, Firatli-Tuglular T, Ozdogu H, Aydogdu I, Konuk N, Sucak G, Kaygusuz I, Karakus S, Kaya E, Ali R, Gulbas Z, Ozet G, Goker H, Undar L. Addition of thalidomide to oral melphalan/prednisone in patients with multiple myeloma not eligible for transplantation: results of a randomized trial from the Turkish Myeloma Study Group. Eur J Haematol. 2011 Jan;86(1):16-22. doi: 10.1111/j.1600-0609.2010.01524.x. Epub 2010 Nov 22. PMID 20942865
- [Background] Fayers PM, Palumbo A, Hulin C, Waage A, Wijermans P, Beksac M, Bringhen S, Mary JY, Gimsing P, Termorshuizen F, Haznedar R, Caravita T, Moreau P, Turesson I, Musto P, Benboubker L, Schaafsma M, Sonneveld P, Facon T; Nordic Myeloma Study Group; Italian Multiple Myeloma Network; Turkish Myeloma Study Group; Hemato-Oncologie voor Volwassenen Nederland; Intergroupe Francophone du Myelome; European Myeloma Network. Thalidomide for previously untreated elderly patients with multiple myeloma: meta-analysis of 1685 individual patient data from 6 randomized clinical trials. Blood. 2011 Aug 4;118(5):1239-47. doi: 10.1182/blood-2011-03-341669. Epub 2011 Jun 13. PMID 21670471
- [Background] Morgan GJ, Davies FE, Gregory WM, Russell NH, Bell SE, Szubert AJ, Navarro Coy N, Cook G, Feyler S, Byrne JL, Roddie H, Rudin C, Drayson MT, Owen RG, Ross FM, Jackson GH, Child JA; NCRI Haematological Oncology Study Group. Cyclophosphamide, thalidomide, and dexamethasone (CTD) as initial therapy for patients with multiple myeloma unsuitable for autologous transplantation. Blood. 2011 Aug 4;118(5):1231-8. doi: 10.1182/blood-2011-02-338665. Epub 2011 Jun 7. PMID 21652683
- [Background] San Miguel JF, Schlag R, Khuageva NK, Dimopoulos MA, Shpilberg O, Kropff M, Spicka I, Petrucci MT, Palumbo A, Samoilova OS, Dmoszynska A, Abdulkadyrov KM, Schots R, Jiang B, Mateos MV, Anderson KC, Esseltine DL, Liu K, Cakana A, van de Velde H, Richardson PG; VISTA Trial Investigators. Bortezomib plus melphalan and prednisone for initial treatment of multiple myeloma. N Engl J Med. 2008 Aug 28;359(9):906-17. doi: 10.1056/NEJMoa0801479. PMID 18753647
- [Background] Bringhen S, Larocca A, Rossi D, Cavalli M, Genuardi M, Ria R, Gentili S, Patriarca F, Nozzoli C, Levi A, Guglielmelli T, Benevolo G, Callea V, Rizzo V, Cangialosi C, Musto P, De Rosa L, Liberati AM, Grasso M, Falcone AP, Evangelista A, Cavo M, Gaidano G, Boccadoro M, Palumbo A. Efficacy and safety of once-weekly bortezomib in multiple myeloma patients. Blood. 2010 Dec 2;116(23):4745-53. doi: 10.1182/blood-2010-07-294983. Epub 2010 Aug 31. PMID 20807892
- [Background] Palumbo A, Chanan-Khan A, Weisel K, Nooka AK, Masszi T, Beksac M, Spicka I, Hungria V, Munder M, Mateos MV, Mark TM, Qi M, Schecter J, Amin H, Qin X, Deraedt W, Ahmadi T, Spencer A, Sonneveld P; CASTOR Investigators. Daratumumab, Bortezomib, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Aug 25;375(8):754-66. doi: 10.1056/NEJMoa1606038. PMID 27557302
- [Background] Reeder CB, Reece DE, Kukreti V, Chen C, Trudel S, Laumann K, Hentz J, Pirooz NA, Piza JG, Tiedemann R, Mikhael JR, Bergsagel PL, Leis JF, Fonseca R, Stewart AK. Once- versus twice-weekly bortezomib induction therapy with CyBorD in newly diagnosed multiple myeloma. Blood. 2010 Apr 22;115(16):3416-7. doi: 10.1182/blood-2010-02-271676. No abstract available. PMID 20413666
- [Background] Mateos MV, Dimopoulos MA, Cavo M, Suzuki K, Jakubowiak A, Knop S, Doyen C, Lucio P, Nagy Z, Kaplan P, Pour L, Cook M, Grosicki S, Crepaldi A, Liberati AM, Campbell P, Shelekhova T, Yoon SS, Iosava G, Fujisaki T, Garg M, Chiu C, Wang J, Carson R, Crist W, Deraedt W, Nguyen H, Qi M, San-Miguel J; ALCYONE Trial Investigators. Daratumumab plus Bortezomib, Melphalan, and Prednisone for Untreated Myeloma. N Engl J Med. 2018 Feb 8;378(6):518-528. doi: 10.1056/NEJMoa1714678. Epub 2017 Dec 12. PMID 29231133

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03992170/Prot_SAP_000.pdf